CLINICAL TRIAL: NCT03676361
Title: To Evaluate the Renal Tubular Function Pre and Post Nephrectomy in Living Donors
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not initiated
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Pooja Budhiraja, MD, Assistant Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00142279
Record Dates: First submitted 2018-09-10; First posted 2018-09-18 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Kidney Damage
Keywords: Kidney Damage
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Desmopressin (Experimental): All ten subjects will be evaluated pre and post nephrectomy at 6 months.
  Interventions: Drug: Desmopressin

INTERVENTIONS:
Drug: Desmopressin — Subjects will complete a water deprivation test using desmopressin to aid in the determination of maximum tubular concentration capacity before and six months after uni-nephrectomy.

SUMMARY:
The overall goals of this study are to demonstrate the change in renal tubular function in living donors pre and post nephrectomy at 6 months.

DETAILED DESCRIPTION:
The physiologic sequelae of living kidney donation are still poorly understood. Uni-nephrectomy from donation results in decreased number of glomeruli and research has shown that there is glomerular hyperfiltration and glomerular hypertrophy. Uni-nephrectomy also results in a decreased number of tubules, but there is not much data about possible tubular injury post donation and its long term effects on donors.

Our overall hypothesis is that post uni-nephrectomy tubular function, measured by maximum urine concentration capacity, will be decreased and may be a more sensitive marker of kidney damage than standard tests, such as urine albumin, serum creatinine, estimated glomerular filtration rate (eGFR), or measured urine creatinine clearance (CrCl). The goal of this study is to evaluate the effect of uni-nephrectomy on renal tubular function and its potential in being an early and more sensitive marker in kidney injury when compared to standard tests.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years of age, who has been evaluated and approved as a potential living donor by the multi-disciplinary committee. All donors undergo a standard medical, social, and psychological pre- donation assessment
* Only patients who are able to sign their own consent form may be included in this study.
* Subjects must be able and willing, in the investigator's opinion, to complete all study requirements.

Exclusion Criteria:

* Subjects denied for donation for any medical, social or surgical reason to be living donor.
* Patients who are contraindicated or relatively contraindicated for DDAVP: a. patients with von Willebrand disease; b. Patients with habitual or psychogenic polydipsia; c. Patients with coronary artery insufficiency and/or hypertensive cardiovascular disease; d. Patients with conditions associated with fluid and electrolyte imbalance, such as cystic fibrosis, heart failure, and renal disorders; e. Patients predisposed to thrombus formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Percentage change in tubular function (urine osmolality measured in MOSMOL/K) pre and post nephrectomy as assessed through water deprivation and administration of desmopressin. | 6 months
  Tubular function is measured as maximal urine concentrating capacity reached after water deprivation and administration of desmopressin.

SECONDARY OUTCOMES:
Sensitivity of serum creatinine when compared to change in tubular function, pre and post nephrectomy as measured in MG/DL. | 6 months
  To test correlations between biomarkers all variables will be log-normalized and Pearson's regression analysis will be used
Sensitivity of urine albumin excretion when compared to change in tubular function, pre and post nephrectomy as measured in MCG/ML. | 6 months
  To test correlations between biomarkers all variables will be log-normalized and Pearson's regression analysis will be used
Sensitivity of eGFR when compared to change in tubular function, pre and post nephrectomy as measured in mL/min. | 6 months
  To test correlations between biomarkers all variables will be log-normalized and Pearson's regression analysis will be used

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Budhiraja, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States